CLINICAL TRIAL: NCT05982457
Title: The Effect of Virtual Reality Application in Cervical Dilatation and Effacement Teaching on Students' Satisfaction, Self-Confidence and Anxiety Levels
Brief Title: The Effect of Virtual Reality Application in Cervical Dilatation and Effacement Teaching
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sevgi Beyazgül (Other)
Responsible Party: Sponsor-Investigator, Sevgi Beyazgül, midwife, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023/74
Record Dates: First submitted 2023-07-12; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Virtual Reality; Educational
Keywords: cervical dilation; midwifery education; simulation; virtual reality

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality group (Experimental): After the introduction and information is given, the lens and pupil distances of the virtual reality glasses will be adjusted according to each student and the students will be provided to wear them. The application will be made one-on-one with each student. The application will be carried out sitting in the laboratory. While the students are inside the application, the interface will be introduced through the images projected to the computer simultaneously. Cervical dilatation and effacement application will be watched using virtual glasses. Then, the students will be asked to use their hands to touch the perineum of the woman and make the image transparent, and it will be ensured that they watch the cervix structures again. Each student will use the virtual glasses for an average of 20-25 minutes.
  Interventions: Behavioral: virtual reality group
- Model group (No Intervention): After the introduction and briefing, the students will be provided to perform cervical dilatation and effacement application on the model in accordance with the Cervical Dilatation and Effacement Learning Guide with each student in the laboratory environment.

INTERVENTIONS:
Behavioral: virtual reality group — Before the training, the Descriptive Information Form and the State and Trait Anxiety Inventory as a pre-test will be applied by face interview method. They will study for two hours. After the introduction and information, the lens and pupil distances of the virtual reality Glasses will be adjusted according to each student and students are expected to wear their vision. The application is the same for every student. Students will be introduced through the images projected to the computer simultaneously while in the application. Cervical dilation and effacement application will be monitored using virtual reality glasses. Next, the students will be asked to touch the woman's perineum with their hands to make her image transparent and we ask them to watch the cervix structures again. After the application, "Learning Satisfaction and Self-Confidence in Learning Scale" and "State and Trait Anxiety Inventory" will be applied as a post-test.
  Arms: virtual reality group

SUMMARY:
The aim of this project is to determine the effect of virtual reality application in cervical dilatation and effacement teaching on students' satisfaction, confidence and anxiety levels.

DETAILED DESCRIPTION:
Midwifery education is extremely important in terms of training midwives specialized in mother-child health. Cervical dilation and effacement is one of the subjects that should be learned well in order to manage the birth process well. Dilatation and effacement of the cervix is the enlargement (dilatation) and thinning (effacement) of the cervical opening and cervical canal when labor begins. Cervical dilation and effacement training is a tactile skill practice that requires constant repetition and practice. Therefore, it cannot be learned by observing, effective learning can be achieved by experiencing it repeatedly in pregnant women. Midwifery students gain experience in the teaching process by practicing with simulation training, laboratory studies and clinical applications. When the literature is examined, no study has been found about the virtual reality application related to cervical dilatation and effacement teaching. The study will be an original study as it focuses on the effect of virtual reality application in cervical dilatation and effacement education on students' satisfaction, self-confidence and anxiety levels. The findings of the study will shed light on the literature in terms of determining the effects of virtual reality application on students in cervical dilatation and effacement teaching. In addition, our project will be a pioneering study in terms of the use of virtual reality application in cervical dilatation and effacement teaching. Within the scope of the study, students will be examined in the focus of their satisfaction, self-confidence and anxiety levels. In this respect, the study will increase awareness in terms of revealing the effects of virtual reality application, which is one of the different simulation teaching methods in cervical dilatation and effacement teaching. Students will be examined as part of the study. In this way, students who have not received cervical dilatation and effacement training with virtual reality application before will have the opportunity to evaluate their exposure to this method.

ELIGIBILITY:
Inclusion Criteria:

* Being a third year student of the Midwifery Department,
* Not having received training in cervical dilation and effacement application
* Volunteering to participate in the study

Exclusion Criteria:

* Not voluntarily participating in the study,
* Having received training in cervical dilatation and effacement

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Descriptive Information Form | 5 minutes before the study
  It consists of nine questions questioning students' socio-demographic characteristics, knowledge of cervical dilatation and effacement, and their virtual reality application experiences.

SECONDARY OUTCOMES:
Student Satisfaction and Self-Confidence in Learning Scale | 5 minutes after the study
  In the sub-dimension of satisfaction with learning; In the sub-dimension of self-confidence, five items measuring satisfaction with the teaching method, variety of learning materials, facilitation, motivation and the suitability of simulation in general; The content adequacy includes eight items: self-confidence, content requirement, skill development, available resources, and information on how to get help to solve clinical problems in simulation. Responses are scored on a five-point Likert system, ranging from 1 (strongly disagree) to 5 (strongly agree), and the total score varies between 13-65.

OTHER OUTCOMES:
State and Trait Anxiety Inventory | 30 minutes after study
  State-Trait Anxiety Inventory; It consists of a total of 40 items, namely the State Anxiety Scale consisting of 20 items and the Trait Anxiety Scale consisting of 20 items. The State Anxiety Inventory requires individuals to describe how they feel under certain conditions at a certain moment, and to answer the items by taking into account their feelings about the situation they are in.